CLINICAL TRIAL: NCT03014258
Title: A Systems Biology Approach to Malaria Immunity: Repetitive Controlled Human Malaria Infection (CHMI) Study in Malaria-Naïve Adults Using NF54 Strain Plasmodium Falciparum (Pf)
Brief Title: A Systems Biology Approach to Malaria Immunity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15-0058
Record Dates: First submitted 2016-12-15; First posted 2017-01-09 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05-27

CONDITIONS: Plasmodium Falciparum Infection
Keywords: Biology; falciparum; Immunity; Infections; Malaria; Pf; Plasmodium; Systems
MeSH Terms: conditions — Infections; Malaria

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control Cohort 1 (Active Comparator): Immunologic malaria-naïve subjects will undergo CHMI #2 with 5 NF54 P. falciparum-infected mosquitoes at months 8-9. n=6.
  Interventions: Biological: NF54 P. falciparum malaria challenge
- Control Cohort 2 (Active Comparator): Immunologic malaria-naïve subjects will undergo a CHMI #3 with 5 NF54 P. falciparum-infected mosquitoes at 6-12 months post CHMI #2. n=6.
  Interventions: Biological: NF54 P. falciparum malaria challenge
- Control Cohort 3 (Active Comparator): Immunologic malaria-naïve subjects will undergo a CHMI #4 with 5 NF54 P. falciparum-infected mosquitoes at 6-12 months post CHMI #3. n=6.
  Interventions: Biological: NF54 P. falciparum malaria challenge
- Control Cohort 4 (Active Comparator): Immunologic malaria-naïve subjects will undergo a CHMI #5 with 5 NF54 P. falciparum-infected mosquitoes at 6-12 months post CHMI #4. n=6.
  Interventions: Biological: NF54 P. falciparum malaria challenge
- Repeat CHMI (Experimental): Subjects will initially be challenged with 5 uninfected mosquitoes (mock), followed by 5 challenges (CHMI # 1-5) with 5 NF54 P. falciparum-infected mosquitoes 2, 8, 14-20, and 20-32, and 32-36 months later. n=10.
  Interventions: Biological: NF54 P. falciparum malaria challenge

INTERVENTIONS:
Biological: NF54 P. falciparum malaria challenge — Aseptically-raised A. stephensi female mosquitoes infected with aseptically-raised P. falciparum parasites of the NF54 strain.

SUMMARY:
This is a phase I study that will assess the acquisition of immunity to Pf malaria over the course of 5 sequential Controlled Human Malaria Infections (CHMI) over 2-4 years, in 10 healthy adult participants. 10 subjects will initially be challenged with 5 uninfected mosquitoes (mock), followed by 5 challenges with 5 mosquitoes infected with drug sensitive, P. falciparum parasites (strain NF54) 2, 8, 14-20, 20-32, and 32-36 months later. For the final four infective CMHIs six additional immunologic malaria-naïve subjects will be enrolled and challenged as infectivity controls. If dropouts occur within the original 10 person cohort, and two or more CHMI remain, back-up replacement volunteers will be recruited to undergo successive CHMI with the core group. All volunteers (repeat CHMI subjects and infectivity controls) will be evaluated as part of an inpatient stay (or outpatient daily follow-up) to diagnose Pf malaria infection and treat with Coartem(R) (artemether/lumefantrine) or Malarone(R) (Atovaquone/proguanil). Daily observation will occur from Study Days 9-19 or until three-day directly observed therapy for P. falciparum infection is complete and two negative smears separated by a time interval >12 hours have been documented. A third negative smear >12 hours after the previous two daily smears will be documented to affirm malaria cure. Infectivity Controls enrolled as part of CHMI #5 will be treated based on concomitant us qPCR results. The repeat CHMI subjects will have additional outpatient visits days 1, 3, 5, and 7 after the challenge to obtain blood samples to monitor the development of immunity. The study is expected to last for 48 months and will include approximately 34 healthy male and female volunteers (10 active study volunteers and 18 naïve controls to confirm Pf infectivity during the 2nd -5th CHMI challenges) ages 18 to 50 years, inclusive, from the greater Baltimore community. The primary objective of this study is to determine whether protective immunity against parasite infection develops following repeat CHMI.

DETAILED DESCRIPTION:
This is a phase I study that will assess the acquisition of immunity to Pf malaria over the course of 5 sequential Controlled Human Malaria Infections (CHMI) over 2-4 years, in 10 healthy adult participants. 10 subjects will initially be challenged with 5 uninfected mosquitoes (mock), followed by 5 challenges with 5 mosquitoes infected with drug sensitive, P. falciparum parasites (strain NF54) 2, 8, 14-20, 20-32, and 32-36 months later. For the final four infective CMHIs six additional immunologic malaria-naïve subjects will be enrolled and challenged as infectivity controls. If dropouts occur within the original 10 person cohort, and two or more CHMI remain, back-up replacement volunteers will be recruited to undergo successive CHMI with the core group. All volunteers (repeat CHMI subjects and infectivity controls) will be evaluated as part of an inpatient stay (or outpatient daily follow-up) to diagnose Pf malaria infection and treat with Coartem(R) (artemether/lumefantrine) or Malarone(R) (Atovaquone/proguanil). Daily observation will occur from Study Days 9-19 or until three-day directly observed therapy for P. falciparum infection is complete and two negative smears separated by a time interval >12 hours have been documented. A third negative smear >12 hours after the previous two daily smears will be documented to affirm malaria cure. Infectivity Controls enrolled as part of CHMI #5 will be treated based on concomitant us qPCR results. The repeat CHMI subjects will have additional outpatient visits days 1, 3, 5, and 7 after the challenge to obtain blood samples to monitor the development of immunity. The study is expected to last for 48 months and will include approximately 34 healthy male and female volunteers (10 active study volunteers and 18 naïve controls to confirm Pf infectivity during the 2nd -5th CHMI challenges) ages 18 to 50 years, inclusive, from the greater Baltimore community. The primary objective of this study is to determine whether protective immunity against parasite infection develops following repeat CHMI. The secondary objectives are to: 1) determine whether clinical signs and symptoms of malaria decrease in intensity and duration following repeat CHMI, 2) track the production of antibodies that react with P. falciparum sporozoites and blood stage parasites.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant/non-lactating female between the ages of 18 and 50 years, inclusive.
2. Able and willing to participate for the duration of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to complete the informed consent process.
5. Willing to donate blood for sample storage to be used for future research (Note: refusal to allow future use is exclusionary).
6. Willing to refrain from blood donation to blood banks for 3 years following P. falciparum CHMI.
7. Agrees not to travel to a malaria endemic region during the entire course of study participation.
8. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) = / < 35.

   Laboratory Criteria within 56 days prior to enrollment:
9. Hemoglobin = / >11.2 g/dL for women; = / > 12.6 g/dL for men.
10. Platelet count within institutional normal range.
11. Alanine aminotransferase (ALT) = / < upper limit of normal.
12. Serum creatinine = / < upper limit of normal.
13. Negative for HIV and Hepatitis B/C infection.

    Laboratory Criterion documented any time prior to enrollment:
14. Negative sickle cell screening test.

    Female-Specific Criteria:
15. Negative beta-HCG pregnancy test (serum) on day of screening or urine pregnancy test at subsequent time points for women of childbearing potential.
16. Women of childbearing potential (exclusive of women in a same sex relationship) must agree to use effective means of birth control.* *(e.g. oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner). Women with a history of amenorrhea (> 1 year duration) or surgical or chemical sterilization (e.g. tubal ligation, hysterectomy, other) must provide written documentation of infertility from a health care provider.

Exclusion Criteria:

1. Women who are breast-feeding or planning to become pregnant during the time interval needed to complete the study.
2. Receipt of a malaria vaccine in a prior clinical trial.
3. Any history of malaria infection.
4. Evidence of increased cardiovascular disease risk; defined as > 10% five year risk by the non-laboratory method.
5. Current use of systemic immunosuppressant pharmacotherapy.
6. History of a splenectomy, sickle cell disease or sickle cell trait.
7. Known history of anaphylactic response to mosquito-bites; or known allergy to artemether lumefantrine or atovaquone or proguanil or other component of the product.
8. Participation in any study involving investigational vaccine or drug within 4 weeks prior to enrollment, or expects to receive vaccine or drug during the 2-month post-challenge period.
9. Use or planned use of any drug with anti-malarial activity that would coincide with challenge.
10. Anticipated use of medications known to cause drug reactions with atovaquone-proguanil (Malarone(R)) such as cimetidine, metoclopramide, antacids, and kaolin.
11. Plans to undergo surgery (elective or otherwise) between enrollment and 4 weeks (28 days) after any of the challenges.
12. Received a licensed vaccine within 1 month prior to enrollment in this study or expects to receive one during the 28 day post challenge period.
13. History of psychiatric disorders or behavioral tendencies (including active alcohol or drug abuse) that in the opinion of the investigator would make compliance with the protocol difficult.* *Medical and psychiatric illness defined as personality disorders, anxiety disorders, or schizophrenia or social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent or to comply with the protocol schedule.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-07 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects testing positive for parasites | Study Day 6 through Study Day 29
  As measured using real-time quantitative polymerase chain reaction (PCR)
Percentage of subjects with positive malaria smear | Study Day 9 through Study Day 29
  For infectivity controls enrolled into infective CHMI #5, malaria detection will rely upon ultra-sensitive quantitative polymerase chain reaction (us-qPCR) to ensure safety while conducting this portion of the study as an outpatient
Quantification of parasite infection | Study Day 6 through Study Day 29
  As measured using real-time quantitative polymerase chain reaction (PCR) during the surveillance period after infected CHMI.

SECONDARY OUTCOMES:
Antibody reactivity against Circumsporozoite protein (CSP) | Up to Study Day 21
  Measured using plasma obtained during the surveillance period. Antibody reactivity is defined as the optical density at 410 nM of a 1/300 dilution of the volunteers plasma sample minus the optical density at 410 nM of a 1/300 dilution of the volunteer's baseline sample.
Antibody reactivity against Glutamate-rich protein (GLURP) | Up to Study Day 21
  Measured using plasma obtained during the surveillance period. Antibody reactivity is defined as the optical density at 410 nM of a 1/300 dilution of the volunteers plasma sample minus the optical density at 410 nM of a 1/300 dilution of the volunteer's baseline sample.
Antibody reactivity against Plasmodium Falciparum liver- and erythrocytic-stage antigen | Up to Study Day 21
  Measured using plasma obtained during the surveillance period. Antibody reactivity is defined as the optical density at 410 nM of a 1/300 dilution of the volunteers plasma sample minus the optical density at 410 nM of a 1/300 dilution of the volunteer's baseline sample.
Antibody reactivity against Plasmodium Falciparum pre-erythrocytic antigen | Up to Study Day 21
  Measured using plasma obtained during the surveillance period. Antibody reactivity is defined as the optical density at 410 nM of a 1/300 dilution of the volunteers plasma sample minus the optical density at 410 nM of a 1/300 dilution of the volunteer's baseline sample.
Percentage of subjects displaying signs and symptoms attributable to malaria | Study Day 6 through Study Day 29
  Such as malaise, chills/rigors, nausea, vomiting, dizziness, arthralgia, abdominal pain, myalgia, and headache
Percentage of subjects with fever attributable to malaria | Study Day 6 through Study Day 29
  Fever as defined as >38 degrees Celsius

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ferrer P, Berry AA, Bucsan AN, Prajapati SK, Krishnan K, Barbeau MC, Rickert DM, Guerrero SM, Usui M, Abebe Y, Patil A, Chakravarty S, Billingsley PF, Pa'ahana-Brown F, Strauss K, Shrestha B, Nomicos E, Deye GA, Sim BKL, Hoffman SL, Williamson KC, Lyke KE. Repeat controlled human Plasmodium falciparum infections delay bloodstream patency and reduce symptoms. Nat Commun. 2024 Jun 18;15(1):5194. doi: 10.1038/s41467-024-49041-2. PMID 38890271